CLINICAL TRIAL: NCT02501330
Title: DRUG USE INVESTIGATION OF BOSUTINIB FOR CML (POST MARKETING COMMITMENT PLAN)
Brief Title: Safety And Efficacy Of Bosutinib
Acronym: BLF
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1871036
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Drug use investigation in Japan
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bosutinib
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — The recommended adult dose of bosutinib is 500 mg orally once daily with food. For newly-diagnosed chronic phase CML, the recommended dose is 400 mg. The dose may be adjusted appropriately according to the patient's condition; however, the maximum dose is 600 mg once daily.
  Other Names: BOSULIF

SUMMARY:
The objective of this surveillance is to collect information about

1. adverse drug reaction not expected from the LPD (unknown adverse drug reaction)
2. the incidence of adverse drug reactions in this surveillance
3. factors considered to affect the safety and/or efficacy of this drug.

DETAILED DESCRIPTION:
The patients should be registered by central registration system.

ELIGIBILITY:
Inclusion Criteria:

* Chronic myelogenous leukemia patients resistant or intolerant to prior treatment there is no experience with this drug
* Newly-diagnosed chronic phase Chronic myelogenous leukemia patients there is no experience with this drug

Exclusion Criteria:

* Patients with a history of hypersensitivity
* Women who may possibly be pregnant or become pregnant

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who have been treated with Bosutinib
Sampling Method: Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse drug reactions | 24 weeks
Cytogenetic response | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Shibuya-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871036&StudyName=Drug%20Use%20Investigation%20Of%20Bosutinib%20For%20Cml%20%28post%20Marketing%20Commitment%20Plan%29